CLINICAL TRIAL: NCT03794648
Title: The Feasibility and Preliminary Efficacy of a Mobile Interactive Supervised Therapy (MIST) Intervention for Improving Medication Adherence of Patients With HIV Infection: a Pilot Randomised Controlled Trial
Brief Title: The Effectiveness of a Mobile Interactive Supervised Therapy (MIST) Intervention for Improving Adherence to HIV Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/00150
Record Dates: First submitted 2018-09-13; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: HIV-infection/Aids
Keywords: mobile app; HIV-infections; medication adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Mobile Interactive Supervised Therapy (MIST)
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Mobile Interactive Supervised Therapy (MIST) — MIST system will send a reminder notification (via push or SMS) to participants 10 to 15 minutes before the scheduled time for taking their medication. Participants will then activate the recording function of the MIST app on their phone, and record themselves taking their medication.Participants will be asked to go through a series of steps for recording the video.
  Arms: Intervention Group

SUMMARY:
A total of 40 HIV infected patients will be randomly assigned into intervention or control group. Participants in the intervention group will use an smart phone application for two months. Participants will receive reminder notifications and use the app to take and send videos of themselves taking the pill(s), uploaded videos will be centrally reviewed by a study nurse . Control group participants will receive standard care. Antiretroviral Therapy adherence will be measured by self-report, pill count, and smart bottle as well as the App. Participants' perceptions of app using experience will be recorded via face to face interview.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* HIV infection diagnosis confirmed by western blot
* Taking a once daily regimen of HIV medications
* Able to take pills orally
* Willing and able to give informed consent

Exclusion Criteria:

* Inability to operate a smart phone
* Active Tuberculosis infection requiring treatment during study (due to additional challenge posed to adherence that may confound the assessment of HIV adherence)
* Substance use
* Visual or hearing impairment
* Cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from one month percentage ART adherence at two months (by MEMScap) | one-month follow-up and two-month follow-up visits
  Change percentage ART adherence over the 2 month study period, as measured by MEMScaps, collected at the 1 and 2 month visits.

SECONDARY OUTCOMES:
Percentage ART adherence (self-reported) | Baseline visit, one-month follow-up visit and two-month follow-up visits (end of study visit)
  Percentage self-reported adherence over a 21 day period (summation of the 7 days preceding each study visit) as measured by a standardised questionnaire at each study visit
Percentage ART adherence (by pill count) | One-month follow-up visit, two-month follow-up visit(end of study visit)
  Percentage adherence over the 2 month study period, as measured by pill count, collected at month 1 and 2 follow-up visits
Variability in time (minutes) between prescribed pill time and actual dose taken | One-month follow-up visit, two-month follow-up visit(end of study visit)
  Variability in time (minutes) between prescribed pill time and actual dose taken, as measured by MEMScaps, collected at the 1 and 2 month visits.
Participants' perceptions on using MIST intervention | two-month follow-up visit (end of the study visit)
  Participants' perception of MIST intervention , assessed at the 2 month visit by a sei-structured interview. The interview mainly addressed five areas namely: perception of overall MIST app use experience, perceived usefulness of each feature, strengths and weakness of MIST, interest in continued to use MIST for future and recommendations for further improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pang Y, Molton JS, Ooi WT, Paton NI, He HG. Preliminary Effects of a Mobile Interactive Supervised Therapy Intervention on People Living With HIV: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 27;8(3):e15702. doi: 10.2196/15702. PMID 32217500